CLINICAL TRIAL: NCT03166137
Title: Comparative Evaluation of Carbon Dioxide Laser and Cryotherapy by Dermoscopy in Treatment of Viral Wart
Brief Title: Carbon Dioxide Laser and Cryotherapy in Treatment of Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kadija Yousef Badawy, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laser,Cryotherapy,Wart
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Common Warts
Keywords: Warts,Laser,Cryotherapy
MeSH Terms: conditions — Warts | interventions — Lasers, Gas; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon dioxide laser group (Experimental): (group A): thirty patients will be treated by application of carbon dioxide laser.
  Interventions: Device: Carbon dioxide laser
- Cryotherapy group (Active Comparator): (group B): thirty patients will be treated by cryotherapy application.
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Carbon dioxide laser — Radiation by carbon dioxide laser
  Arms: Carbon dioxide laser group
Device: Cryotherapy — Device using cooling effect
  Arms: Cryotherapy group

SUMMARY:
Viral warts are common skin conditions seen in both children and adults. Human papilloma virus is responsible for verrucae. Cutaneous manifestation of the human papillomavirus, are extremely common particularly on the hands and feet. Warts can induce hard, thickened skin, black pinpoints, pain or tenderness with significant morbidity for the patients.

DETAILED DESCRIPTION:
A range of types of wart have been identified, varying in shape and site affected, as well as the type of human papillomavirus involved.

These include:

* Common wart (Verruca vulgaris).
* Flat wart (Verruca plana).
* Filiform or digitate wart.
* Genital wart (venereal wart, Condyloma acuminatum, Verruca acuminata).
* Mosaic wart.
* Periungual wart.
* Plantar wart (verruca, Verruca plantaris). Despite the presence of several therapeutic options, treatment of warts can present a challenge and they are not uniformly effective. Viral warts often disappear without treatment. In case of pain, discomfort and long duration they can be treated . Treatment options include cryotherapy, electrocautery, salicylic acid, immune therapy, minor surgery or laser surgery.

Common warts have a distinctive appearance and can usually be diagnosed with the unaided eye; however, early growth stages and post-treatment warts are less easily diagnosed. Published dermoscopic features of common warts include frogspawn pattern, mosaic pattern and dotted, linear, globular or coiled vessels. Mosaic pattern consists of relatively flattened, rounded structures of similar size, resembling a jigsaw puzzle. Frogspawn pattern consists of densely packed papillae, each containing red dot or loop, surrounded by a whitish halo. Vascular structures seen dermoscopically in common warts as red or black dotted, linear, globular and coiled vessels. Haemorrhages are possible additional features, with black dots corresponding to thrombosed vessels. Hairpin vessels were usually seen in non-wart lesions.

In this study, we aim to compare two therapeutic modalities, the clinical effectiveness and safety of carbon dioxide laser and cryotherapy in the treatment of viral warts together with dermoscopic evaluation of viral warts before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with common warts male or females any age.
2. Patient is able to read and understand English and will give written informed consent to participate.
3. Patient elects to undergo carbon dioxide laser therapy or cryotherapy for treatment of common warts.
4. Warts to be treated will be located only on the hands.

Exclusion Criteria:

1. Non cooperative patients.
2. Patients on other lines of treatment.
3. Pregnant and lactating females.
4. Patients receiving topical treatment in the previous two weeks.
5. Secondary infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Number and size of the lesions. | Two months
  Dermoscopic evaluation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vlahovic TC, Khan MT. The Human Papillomavirus and Its Role in Plantar Warts: A Comprehensive Review of Diagnosis and Management. Clin Podiatr Med Surg. 2016 Jul;33(3):337-53. doi: 10.1016/j.cpm.2016.02.003. Epub 2016 Mar 29. PMID 27215155
- [Result] Kwok CS, Gibbs S, Bennett C, Holland R, Abbott R. Topical treatments for cutaneous warts. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD001781. doi: 10.1002/14651858.CD001781.pub3. PMID 22972052
- [Result] Andrews MD. Cryosurgery for common skin conditions. Am Fam Physician. 2004 May 15;69(10):2365-72. PMID 15168956
- [Result] Zalaudek I, Giacomel J, Cabo H, Di Stefani A, Ferrara G, Hofmann-Wellenhof R, Malvehy J, Puig S, Stolz W, Argenziano G. Entodermoscopy: a new tool for diagnosing skin infections and infestations. Dermatology. 2008;216(1):14-23. doi: 10.1159/000109353. PMID 18032894